CLINICAL TRIAL: NCT06945939
Title: Correlation Between Ultrasound Findings Vs Intraoperative Findings in Syndesmotic Injury in Pott's Fracture Weber b and c
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Mohamed Salah Shehata, Toukh-Alqalyubiyah-Egypt, Benha University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Ankle syndesmotic injury
Record Dates: First submitted 2025-03-13; First posted 2025-04-27 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-03

CONDITIONS: Ankle Syndesmotic Injury Associated With Pott's Fracture
Keywords: Syndesmotic ankle injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Correlation between ultrasound findings vs intraoperative findings in syndesmotic ankle injury (Active Comparator): Correlation between ultrasound findings vs intraoperative findings in syndesmotic injury of Pott's B and c
  Interventions: Procedure: Fixation of Pott's fracture b and c

INTERVENTIONS:
Procedure: Fixation of Pott's fracture b and c — Assessment of syndesmotic injury via X-ray, CT, ultrasound and intraoperative

SUMMARY:
This study aims to assess and compare ultrasound findings, radiographic findings and intraoperative findings in cases of Pott's fractures weber types B and C to evaluate the accuracy of ultrasound in diagnosis of syndesmotic injury.

DETAILED DESCRIPTION:
Ankle fractures are among of the most frequently addressed injuries by orthopedic surgeons. Ankle fractures have an incidence rate about 107-145 per 100000 in adult population. Approximately 10% of these fractures are concomitant with syndesmotic injury. This percentage is doubled in patients who need open reduction and internal fixation( ORIF).As a result ,it is essential for orthopedic surgeons to accurately diagnose these injuries,which ocurr in up to 40% of weber type B pott's fracture and up to 80% in pott's c. Failure to properly diagnose or treat these injuries can lead to persistent ankle pain ,functional instability and early osteoarthritis. The ankle joint is a synovial joint that connects leg bones :the fibula which ends distally with lateral malleolus and the tibia which ends distally with tibial plafond , medial malleolus and posterior malleolus ,with the talus.It is a complex hinge joint.) 2.Kennedy JG, Soffe KE, Dalla Vedova P, Stephens MM, O'Brien T, Walsh MG, McManus F( Ankle syndesmosis injuries are common, but diagnosing and treating them can be challenging, often leading to differing opinions among healthcare providers. It is crucial for orthopedic surgeons to recognize the complex nature of these injuries, especially when they involve damage to the interosseous membrane. Patients may seek medical attention years after the initial injury, reporting gradual, worsening pain and swelling following physical activity. These symptoms can significantly affect their quality of life.

Diagnostic dilemma of syndesmotic injury in ankle fracture:

The are different modalities regarding the diagnosis:

* X-ray imaging is one of the most commonly used methods for diagnosing ankle syndesmosis injuries. In a normal anteroposterior radiograph, the tibiofibular overlap should be greater than 6 mm, while in a mortise radiograph, it should exceed 1 mm when measured 1 cm above the tibial plafond. Similarly, the tibiofibular clear space should be less than 6 mm in both anteroposterior and mortise views at the same level. Additionally, the medial clear space should be equal to or less than the distance between the talar dome and the tibial plafond. A reduction in tibiofibular overlap, an increase in tibiofibular clear space, or an increase in medial clear space whether observed on weight-bearing or non weight-bearing radiographs suggests syndesmotic disruption.) 6. Pogliacomi F, De Filippo M, Casalini D, Longhi A, Tacci F, Perotta R, Pagnini F, Tocco S, Ceccarelli( While standard radiographic views are useful for evaluating moderate-to-severe ankle syndesmosis injuries, detecting subtle syndesmotic widening remains challenging.
* Computed tomography (CT) provides a clear and direct visualization of the positional alignment of the distal tibiofibular syndesmosis. It allows precise measurement of the syndesmotic gap and facilitates comparison with the contralateral side. As a result, CT is particularly valuable for diagnosing ankle syndesmosis injuries when radiographic findings are inconclusive. A syndesmosis injury is generally indicated if the gap exceeds 6 mm or is more than 2 mm wider than the opposite side.Exposure to CT radiation can cause many hazards to patients.) 3.Elgafy H, Semaan HB, Blessinger B, Wassef A, Ebraheim NA(.
* MRI is the preferred method for diagnosing syndesmosis injuries due to its high sensitivity and specificity. However, examination techniques particularly slice orientation and ankle positioning require standardization to ensure optimal visualization of the distal tibiofibular ligament. The oblique orientation of ligament fibers may result in false positives when compared to intraoperative findings. Additional associated injuries, such as anterior talofibular ligament tears, bone edema, osteochondral lesions, or distal tibiofibular joint incongruities, may also be present. These findings can include ligament discontinuity or irregular, curved, or indistinct ligament contours.The high cost and non availability of MRI hinder and limit it's use in clinical practice.) 8.Kellett JJ, Lovell GA, Eriksen DA, Sampson MJ. Diagnostic imaging of ankle syndesmosis injuries:(
* Ultrasound offers a cost-effective and readily available option that could serve as a screening tool for syndesmotic ligamentous injuries in the ankle. The ultrasound evaluation begins by examining the anterior compartment to check for joint fluid, synovitis, and osteophytes on the tibia or talus. Tendons in the extensor, medial, and lateral compartments are evaluated in both longitudinal and transverse planes. The lateral compartment assessment focuses on the anterior talofibular ligament (ATFL) and calcaneofibular ligament (CFL). In the medial compartment, the deltoid ligament is assessed in the oblique coronal plane. The syndesmosis is imaged in all cases using the transverse plane through an anterior approach. The anterior-inferior tibiofibular ligament (AITFL) is inspected for continuity and contour, and the tibia-fibula distance (clear space) is measured.) 1.Hagemeijer NC, Lubberts B, Saengsin J, Bhimani R, Sato G, Waryasz GR, Kerkhoffs GMMJ, DiGiovanni CW, Guss D(

ELIGIBILITY:
Inclusion Criteria:

* Patients who will present at Benha university hospitals with ankle fractures weber type B,B/C and C. Patients will be enrolled in the study as long as they are generally fit for the operation and their functional requirements justify the procedure.The study will include only patients older than 18years old with closed fractures once their skin condition allows.

Exclusion Criteria:

* Age less than 18y and more than 60yr.
* Previous history of ipsilateral ankle fracture or fixation.
* History of chronic ankle ankle instability or recurrent ankle sprains.
* significant ankle or subtalar osteoarthritis.
* Pathological ankle fracture .
* Patients with open ankle fracture.
* Patients with ankle fracture with vascular injury or neurological impairment.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-04-15 (Estimated); Primary Completion 2026-04-15 (Estimated); Study Completion 2026-05-15 (Estimated)

PRIMARY OUTCOMES:
Syndesmotic ankle injury in pott's fracture | baseline
  Correlation between :1-ultrasound findings regarding syndesmotic injury in pott's fracture weber b and c:*AITFL (anterior inferior tibiofibular ligament)for continuity, contour and presence of hematoma.
  * PITFL(posterior inferior tibiofibular ligament) integrity.
  * Deltoid ligament integrity.
  * Measurement of tibiofibular clear space.
  * Measurement of Medial clear space. The transducer (LOGIQ P9-Linear transducer 8/15MH) positioned transverse1cm above ankle joint, where ligament is at its thickness.
Syndesmotic ankle injury in pott's fracture | baseline
  Intraoperative findings in pott's Weber b and c fracture guided with guided with arthroscopy and ORIF (open reduction and internal fixation).
Ankle syndesmotic injury in pott's fracture | baseline
  Preoperative X-ray and CT scanning

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Swords M, Brilhault J, Sands A. Acute and Chronic Syndesmotic Injury: The Authors' Approach to Treatment. Foot Ankle Clin. 2018 Dec;23(4):625-637. doi: 10.1016/j.fcl.2018.07.007. Epub 2018 Sep 24. PMID 30414657
- [Background] Fort NM, Aiyer AA, Kaplan JR, Smyth NA, Kadakia AR. Management of acute injuries of the tibiofibular syndesmosis. Eur J Orthop Surg Traumatol. 2017 May;27(4):449-459. doi: 10.1007/s00590-017-1956-2. Epub 2017 Apr 8. PMID 28391516
- [Background] Kellett JJ, Lovell GA, Eriksen DA, Sampson MJ. Diagnostic imaging of ankle syndesmosis injuries: A general review. J Med Imaging Radiat Oncol. 2018 Apr;62(2):159-168. doi: 10.1111/1754-9485.12708. Epub 2018 Feb 5. PMID 29399975
- [Background] Akoh CC, Phisitkul P. Anatomic Ligament Repairs of Syndesmotic Injuries. Orthop Clin North Am. 2019 Jul;50(3):401-414. doi: 10.1016/j.ocl.2019.02.004. Epub 2019 Apr 16. PMID 31084843
- [Background] Shoji H, Teramoto A, Murahashi Y, Watanabe K, Yamashita T. Syndesmotic instability can be assessed by measuring the distance between the tibia and the fibula using an ultrasound without stress: a cadaver study. BMC Musculoskelet Disord. 2022 Mar 18;23(1):261. doi: 10.1186/s12891-022-05221-z. PMID 35303853
- [Background] Pogliacomi F, De Filippo M, Casalini D, Longhi A, Tacci F, Perotta R, Pagnini F, Tocco S, Ceccarelli F. Acute syndesmotic injuries in ankle fractures: From diagnosis to treatment and current concepts. World J Orthop. 2021 May 18;12(5):270-291. doi: 10.5312/wjo.v12.i5.270. eCollection 2021 May 18. PMID 34055585
- [Background] Hagemeijer NC, Saengsin J, Chang SH, Waryasz GR, Kerkhoffs GMMJ, Guss D, DiGiovanni CW. Diagnosing syndesmotic instability with dynamic ultrasound - establishing the natural variations in normal motion. Injury. 2020 Nov;51(11):2703-2709. doi: 10.1016/j.injury.2020.07.060. Epub 2020 Jul 27. PMID 32741605
- [Background] Baltes TPA, Arnaiz J, Geertsema L, Geertsema C, D'Hooghe P, Kerkhoffs GMMJ, Tol JL. Diagnostic value of ultrasonography in acute lateral and syndesmotic ligamentous ankle injuries. Eur Radiol. 2021 Apr;31(4):2610-2620. doi: 10.1007/s00330-020-07305-7. Epub 2020 Oct 7. PMID 33026501
- [Background] Elgafy H, Semaan HB, Blessinger B, Wassef A, Ebraheim NA. Computed tomography of normal distal tibiofibular syndesmosis. Skeletal Radiol. 2010 Jun;39(6):559-64. doi: 10.1007/s00256-009-0809-4. Epub 2009 Oct 15. PMID 19830423
- [Background] Kennedy JG, Soffe KE, Dalla Vedova P, Stephens MM, O'Brien T, Walsh MG, McManus F. Evaluation of the syndesmotic screw in low Weber C ankle fractures. J Orthop Trauma. 2000 Jun-Jul;14(5):359-66. doi: 10.1097/00005131-200006000-00010. PMID 10926245
- [Background] Hagemeijer NC, Lubberts B, Saengsin J, Bhimani R, Sato G, Waryasz GR, Kerkhoffs GMMJ, DiGiovanni CW, Guss D. Portable dynamic ultrasonography is a useful tool for the evaluation of suspected syndesmotic instability: a cadaveric study. Knee Surg Sports Traumatol Arthrosc. 2023 May;31(5):1986-1993. doi: 10.1007/s00167-022-07058-4. Epub 2022 Jul 26. PMID 35881148